CLINICAL TRIAL: NCT00973362
Title: Clinical Evaluation of the APTIMA® HPV Assay on the TIGRIS® DTS® System in Women With ASC-US Pap Test Results and in Women 30 Years of Age or Older With Negative Pap Test Results Using ThinPrep Pap Test Specimens
Brief Title: Clinical Evaluation of the APTIMA® HPV Assay Using the TIGRIS® System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2007HPVASCUS30
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Human Papillomavirus Infection
Keywords: Cervix Cancer; Cervical Intraepithelial Neoplasia (CIN); Human Papillomavirus Virus (HPV); APTIMA HPV Assay; FDA-Approved HPV DNA Test; TIGRIS DTS (direct tube sampling) System; Clinical Sensitivity (%); Clinical Specificity (%); Positive Predictive Value [PPV] (%); Negative Predictive Value [NPV] (%); Atypical Squamous Cells Undetermined Significance (ASC-US); Relative Risk
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Atypical Squamous Cells of the Cervix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjunct (i.e. Normal Pap) (Other): The Adjunct study will evaluate APTIMA HPV Assay clinical performance for detecting high-risk HPV types in female subjects 30+ years of age with negative (NILM) cytology results from routine Pap testing. This will be accomplished by evaluating the assay performance compared to known cervical disease status at baseline and after a 3-year follow-up period. A comparator FDA-Approved HPV DNA test is reported.
  Interventions: Device: APTIMA HPV Assay; Device: FDA-Approved HPV DNA Test
- ASC-US (Other): The ASC-US study will evaluate the APTIMA HPV Assay clinical performance for detecting high-risk HPV types in subjects with ASC-US Pap test results from routine Pap testing and known cervical disease status (based on colposcopic biopsy results). A comparator FDA-Approved HPV DNA test is reported. There is no follow-up period.
  Interventions: Device: APTIMA HPV Assay; Device: FDA-Approved HPV DNA Test

INTERVENTIONS:
Device: APTIMA HPV Assay — The APTIMA HPV Assay is an in vitro nucleic acid amplification test (NAAT) that qualitatively detects human papillomavirus (HPV) E6/E7 messenger RNA (mRNA) from 14 HPV types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) that are associated with cervical cancer ("high-risk types"). The assay cannot determine the specific high-risk HPV type(s) present and does not cross-react with 5 HPV types that are considered non-oncogenic (not associated with cervical cancer; types 6, 11, 42, 43, and 44).
Device: FDA-Approved HPV DNA Test — A FDA-Approved HPV DNA Test is used as the comparator assay.

SUMMARY:
The purpose of this study is to provide data on the performance of the APTIMA HPV Assay using the TIGRIS System in detecting HPV types that may cause cervical cancer.

DETAILED DESCRIPTION:
The primary objective of the clinical trial is to evaluate the APTIMA HPV Assay, using the TIGRIS System, in cervical cancer screening programs. This will be achieved by determining the performance of the assay for detecting high-risk human papillomavirus (HPV) types in women with known cervical disease status. The assay will be evaluated in sample populations of women with ASC-US Pap test results ("ASC-US results") and women 30 years of age or older ("30+ years of age") with negative (NILM) cytology results.

ELIGIBILITY:
Inclusion Criteria:

* Female 21 years or older (ASC-US study only)
* Female 30 years or older (Adjunct and ASC-US studies)
* Subject attending a participating clinic and undergoing a Pap screening exam during the clinic visit
* Ability to comprehend and sign an IRB-approved Informed Consent Form

Exclusion Criteria:

* Diagnosis of cervical disease (cancer or precancerous condition) in the past 12 months
* Abnormal Pap test result in the past 12 months
* Subject under 18 years of age and consenting to the study without the presence of their parent or legal guardian
* Known to be pregnant
* Having an illness or medical condition that could interfere with or affect the conduct, results, and/or completion of the clinical trial
* Having an illness or medical condition that the investigator or physician feels would create an unacceptable risk to the subject if she enrolled into the clinical trial
* Prior vaccination for HPV

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12896 (Actual)
Dates: Start 2008-03; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reid, PhD, Study Director — Gen-Probe, Incorporated
Locations (17):
- United States (17):
  - NEA Clinic Women's Clinic, Jonesboro, Arkansas
  - San Fernando Valley Research, Canoga Park, California
  - Healthcare Partners of Monterey Park, Los Angeles, California
  - Diverse Research Solutions, Oxnard, California
  - REMEK, Pomona, California
  - West Coast OB-Gyn, San Diego, California
  - HealthCare Partners, Torrance, California
  - Penninsula Research Associates, Torrance, California
  - Community Medical Research of South Florida, Miami, Florida
  - Insignia Clinical Research, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Indiana Univ. School of Medicine Dept of Pathology Wishard Health Sciences, Indianapolis, Indiana
  - Saginaw Valley Medical Research, Saginaw, Michigan
  - PPS Clinical, Chesterfield, Missouri
  - Planned Parenthood of Eastern Arkansas and Oklahoma, Tulsa, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Adams Patterson OB-GYN, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adjunct (i.e. Normal Pap): The Adjunct study will evaluate APTIMA HPV Assay performance for detecting high-risk HPV types in female subjects 30+ years of age with negative (NILM) cytology results from routine Pap testing. This will be accomplished by evaluating the assay performance compared to known cervical disease status at baseline and after a 3-year follow-up period.
  APTIMA HPV Assay: The APTIMA HPV Assay is an in vitro nucleic acid amplification test (NAAT) that qualitatively detects human papillomavirus (HPV) E6/E7 messenger RNA (mRNA) from 14 HPV types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) that are associated with cervical cancer ("high-risk types"). The assay cannot determine the specific high-risk HPV type(s) present and does not cross-react with 5 HPV types that are considered non-oncogenic (not associated with cervical cancer; types 6, 11, 42, 43, and 44).
- ASC-US: The ASC-US study will determine the sensitivity and specificity of the APTIMA HPV Assay for detecting high-risk HPV types in subjects with ASC-US Pap test results from routine Pap testing and known cervical disease status (based on colposcopic biopsy results).
  APTIMA HPV Assay: The APTIMA HPV Assay is an in vitro nucleic acid amplification test (NAAT) that qualitatively detects human papillomavirus (HPV) E6/E7 messenger RNA (mRNA) from 14 HPV types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) that are associated with cervical cancer ("high-risk types"). The assay cannot determine the specific high-risk HPV type(s) present and does not cross-react with 5 HPV types that are considered non-oncogenic (not associated with cervical cancer; types 6, 11, 42, 43, and 44).
  There is no follow-up period for the ASC-US Arm of the study, only for the Adjunct ARM has a three (3) year follow-up period.
Period: Baseline Evaluation
Arm/Group | Adjunct (i.e. Normal Pap) | ASC-US
Started | 11644 | 1252
Evaluable for Analysis | 10871 | 958
Conclusive Disease Status | 819 | 939
Completed | 10871 | 1029
Not Completed | 773 | 223
Not completed — W/D, later determined to be ineligible | 25 | 0
Not completed — No colposcopy visit | 62 | 0
Not completed — Inevaluable | 686 | 223
Period: 3-Year Follow-up
Arm/Group | Adjunct (i.e. Normal Pap) | ASC-US
Started | 10871 | 0 (ASC-US study arm did not have a follow-up period)
Completed | 10854 | 0
Not Completed | 17 | 0
Not completed — Lost to Follow-up | 17 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Evaluable Analysis Population
Groups:
- ASC-US: The ASC-US study will determine the sensitivity and specificity of the APTIMA HPV Assay for detecting high-risk HPV types in subjects with ASC-US Pap test results from routine Pap testing and known cervical disease status (based on colposcopic biopsy results).
  APTIMA HPV Assay: The APTIMA HPV Assay is an in vitro nucleic acid amplification test (NAAT) that qualitatively detects human papillomavirus (HPV) E6/E7 messenger RNA (mRNA) from 14 HPV types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) that are associated with cervical cancer ("high-risk types"). The assay cannot determine the specific high-risk HPV type(s) present and does not cross-react with 5 HPV types that are considered non-oncogenic (not associated with cervical cancer; types 6, 11, 42, 43, and 44).
- Total: Total of all reporting groups
Arm/Group | Adjunct (i.e. Normal Pap) | ASC-US | Total
Number analyzed (Participants) | 10871 | 958 | 11829
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (10.1) | 33.8 (10.3) | 43.3 (10.5)
Age, Customized [Number; unit: participants]
  21 - <30 years | 0 | 418 | 418
  30 - <40 years | 4199 | 266 | 4465
  40+ years | 6672 | 274 | 6946
Gender [Count of Participants; unit: Participants]
  Female | 10871 | 958 | 11829
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3421 | 195 | 3616
  Not Hispanic or Latino | 6881 | 712 | 7593
  Unknown or Not Reported | 569 | 51 | 620
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 76 | 12 | 88
  Asian | 622 | 27 | 649
  Native Hawaiian or Other Pacific Islander | 48 | 1 | 49
  Black or African American | 1358 | 218 | 1576
  White | 6831 | 566 | 7397
  More than one race | 128 | 28 | 156
  Unknown or Not Reported | 1808 | 106 | 1914
Region of Enrollment [Number; unit: participants]
  United States | 10871 | 958 | 11829

OUTCOME MEASURES:

1. Primary Outcome: Adjunct Study Arm: Compare Assay Performance for Aptima HPV Assay to a FDA-Approved HPV Assay for Detecting CIN2+
Description: Adjunct 30+ yrs. Population: Aptima HPV Assay Performance for Detecting CIN2+: Compare Clinical Performance of the Aptima HPV Assay to a FDA-Approved HPV Assay for Detecting CIN2+
Time Frame: Baseline Evaluation
Measure: Number; unit: participants
Groups:
- APTIMA HPV Assay: The Adjunct study will evaluate APTIMA HPV Assay clinical performance for detecting high-risk HPV types in female subjects 30+ years of age with negative (NILM) cytology results from routine Pap testing. This will be accomplished by evaluating the assay performance compared to known cervical disease status at baseline and after a 3-year follow-up period.
  APTIMA HPV Assay: The APTIMA HPV Assay is an in vitro nucleic acid amplification test (NAAT) that qualitatively detects human papillomavirus (HPV) E6/E7 messenger RNA (mRNA) from 14 HPV types (types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) that are associated with cervical cancer ("high-risk types"). The assay cannot determine the specific high-risk HPV type(s) present and does not cross-react with 5 HPV types that are considered non-oncogenic (not associated with cervical cancer; types 6, 11, 42, 43, and 44).
Arm/Group | APTIMA HPV Assay
Number analyzed (Participants) | 819
participants
  Assay Positive, CIN2+ | 15
  Assay Negative, CIN2+ | 5
  Assay Positive, No Disease | 299
  Assay Negative, No Disease | 500
Statistical Analysis 1: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Sensitivity (%) = 75.0, 95% CI 2-sided [53.1 to 88.8]
Statistical Analysis 2: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Specificity (%) = 62.6, 95% CI 2-sided [59.2 to 65.9]
Statistical Analysis 3: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Positive Predictive Value [PPV] (%) = 4.8, 95% CI 2-sided [3.4 to 5.8]
Statistical Analysis 4: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Negative Predictive Value [NPV] (%) = 99.0, 95% CI 2-sided [98.1 to 99.6]
Statistical Analysis 5: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Prevalence (%) = 2.4
Statistical Analysis 6: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Relative Risk = 4.8, 95% CI 2-sided [1.8 to 13.1] — The relative risk of CIN2+ is defined as the [ absolute risk of APTIMA HPV (Positive Result) / absolute risk of APTIMA HPV (Negative Result) ]

2. Primary Outcome: Adjunct Study Arm: Compare Assay Performance for FDA-Approved HPV DNA Assay to a FDA-Approved HPV Assay for Detecting CIN2+
Description: Adjunct Study Arm: 30+ yrs. Population: FDA-Approved HPV DNA Assay Performance for Detecting CIN2+: Compare Clinical Performance of the Aptima HPV Assay to a FDA-Approved HPV Assay for Detecting CIN2+
Time Frame: Baseline Evaluation
Population: 18 women with Aptima HPV results did not have FDA-Approved DNA test results due to insufficient volume of the cytology specimen for a N of 801 compared to a N of 819 for the Aptima HPV assay results.
Measure: Number; unit: participants
Groups:
- FDA-Approved DNA Test: A FDA-Approved HPV DNA Test is the comparator assay,
Arm/Group | FDA-Approved DNA Test
Number analyzed (Participants) | 801
participants
  Assay Positive, CIN2+ | 16
  Assay Negative, CIN2+ | 3
  Assay Positive, No Disease | 401
  Assay Negative, No Disease | 381
Statistical Analysis 1: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Sensitivity (%) = 84.2, 95% CI 2-sided [62.4 to 94.5]
Statistical Analysis 2: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Specificity (%) = 48.7, 95% CI 2-sided [45.2 to 52.2]
Statistical Analysis 3: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Positive Predictive Value [PPV] (%) = 3.8, 95% CI 2-sided [2.9 to 4.4]
Statistical Analysis 4: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Negative Predictive Value [NPV] (%) = 99.2, 95% CI 2-sided [98.1 to 99.8]
Statistical Analysis 5: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Prevalence (%) = 2.4
Statistical Analysis 6: Comparison: FDA-Approved DNA Test; Test type: Superiority or Other; Relative Risk = 4.9, 95% CI 2-sided [1.4 to 16.7] — The relative risk of CIN2+ is defined as the [ absolute risk of FDA-Approved HPV DNA Assay (Positive Result) / absolute risk of FDA-Approved HPV DNA Assay (Negative Result) ]

3. Secondary Outcome: ASC-US Study Arm: Aptima HPV Assay Performance for Detecting CIN2+ (All Biopsies)
Description: ASC-US Study Arm: 21+ yrs. Population: Aptima HPV assay performance on Tigris System for detecting CIN2+ (All Biopsies)
Time Frame: Baseline Evaluation
Measure: Number; unit: participants
Groups:
- APTIMA HPV Assay: APTIMA HPV Assay Performed on the Tigris System
- FDA-Approved HPV DNA Test: FDA-Approved HPV DNA Test as Comparator
Arm/Group | APTIMA HPV Assay | FDA-Approved HPV DNA Test
Number analyzed (Participants) | 939 | 865
participants
  Assay Positive, CIN2+ | 79 | 79
  Assay Negative, CIN2+ | 12 | 10
  Assay Positive, No Disease | 315 | 343
  Assay Negative, No Disease | 533 | 433
Statistical Analysis 1: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Sensitivity(%) = 86.8, 95% CI 2-sided [78.4 to 92.3]
Statistical Analysis 2: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Specificty = 62.9, 95% CI 2-sided [59.6 to 66.0]
Statistical Analysis 3: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; PPV = 20.1, 95% CI 2-sided [18.1 to 22.0]
Statistical Analysis 4: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; NPV = 97.8, 95% CI 2-sided [96.5 to 98.8]
Statistical Analysis 5: Comparison: APTIMA HPV Assay; Test type: Superiority or Other; Prevalence (%) = 9.7

4. Secondary Outcome: ASC-US Study Arm: FDA-Approved HPV DNA Assay Performance for Detecting CIN2+ (All Biopsies)
Description: ASC_US Study Arm: 21+ yrs. Population for Detecting CIN2+ (All Biopsies): FDA-Approved HPV DNA Assay
Time Frame: Baseline Evaluation
Population: 74 women with Aptima HPV assay results did not have FDA-Approved HPV DNA test results primarily due to insufficient volume of the cytology specimen for an N of 865 results for the FDA-Approved HPV DNA assay compared to 939 results for the Aptima HPV assay.
Measure: Number; unit: participants
Arm/Group | FDA-Approved HPV DNA Test
Number analyzed (Participants) | 865
participants
  Assay Positive, CIN2+ | 79
  Assay Negative, CIN2+ | 10
  Assay Positive, No Disease | 343
  Assay Negative, No Disease | 433
Statistical Analysis 1: Comparison: FDA-Approved HPV DNA Test; Test type: Superiority or Other; Sensitivity (%) = 88.8, 95% CI 2-sided [80.5 to 93.8]
Statistical Analysis 2: Comparison: FDA-Approved HPV DNA Test; Test type: Superiority or Other; Specificity(%) = 55.8, 95% CI 2-sided [52.3 to 59.3]
Statistical Analysis 3: Comparison: FDA-Approved HPV DNA Test; Test type: Superiority or Other; PPV(%) = 18.7, 95% CI 2-sided [17.0 to 20.4]
Statistical Analysis 4: Comparison: FDA-Approved HPV DNA Test; Test type: Superiority or Other; NPV(%) = 97.7, 95% CI 2-sided [96.2 to 98.8]
Statistical Analysis 5: Comparison: FDA-Approved HPV DNA Test; Test type: Superiority or Other; Prevalence(%) = 10.3

ADVERSE EVENTS:
Time Frame: 5 years
Description: 2 years for recruitment for Adjunct and ACS-US Arms with a 3 years follow-up period for the Adjunct Arm
Arm/Group | Adjunct (i.e. Normal Pap) | ASC-US
Serious Adverse Events (participants affected / at risk) | 0/11644 | 0/1252
Other Adverse Events (participants affected / at risk) | 0/11644 | 0/1252

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less